CLINICAL TRIAL: NCT06595238
Title: A Phase IIb Randomised, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety and Tolerability of AZD6234 in Participants Living With Obesity or Overweight With Comorbidity
Brief Title: A Study in Participants With Obesity or Overweight With at Least One Weight-related Comorbidity
Acronym: APRICUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8750C00004; 2024-514000-13-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity or Overweight
Keywords: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): Dose 1
  Interventions: Drug: AZD6234
- Arm 2 (Experimental): Dose 2
  Interventions: Drug: AZD6234
- Arm 3 (Experimental): Dose 3
  Interventions: Drug: AZD6234
- Arm 4 (Placebo Comparator): Placebo - Dose matched with each Experimental arm
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: AZD6234 — IMP injected subcutaneously, once a week. Unit dose strength as per CSP
  Arms: Arm 1; Arm 2; Arm 3
Drug: Placebo comparator — Placebo matching IMP dose injected subcutaneously, once a week.
  Arms: Arm 4

SUMMARY:
A Phase IIb Randomised, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety and Tolerability of AZD6234 compared with placebo, given once a week as subcutaneous injection for 36 weeks, in male and female participants of at least 18 years of age who are living with obesity (body mass index [BMI] ≥ 30 kg/m2), or overweight (BMI ≥ 27 kg/m2) and at least one weight-related comorbidity

DETAILED DESCRIPTION:
The study will comprise of:

A screening period of maximum 28 days

A treatment period of 36 weeks

A follow up period after last dose of study drug

This study will consist of 4 cohorts. Approximately 231 eligible participants will be randomized to AZD6234 or placebo

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* BMI of (a) ≥ 30 kg/m2, or (b) ≥ 27kg/m2 and have a current diagnosis of at least 1 weight-related comorbidities (treated or untreated)
* A stable body weight for 3 months prior to Screening (±5% body weight change)

Exclusion Criteria:

* Have obesity induced by other endocrine disorders, such as Cushing's syndrome or Prader-Willi syndrome
* Has received prescription or non-prescription medication for weight loss within the last 3 months prior to Screening
* Previous or planned (within study period) bariatric surgery or fitting of a weight loss device (eg, gastric balloon or duodenal barrier)
* History of type 1 diabetes mellitus or T2DM

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Percent change in body weight from baseline to week 26 | 26 weeks
  To determine whether AZD6234 is superior to placebo for weight loss
Weight loss ≥ 5% from baseline weight to week 26 | 26 weeks
  To determine whether AZD6234 is superior to placebo in participants with weight loss ≥ 5% from baseline

SECONDARY OUTCOMES:
Weight loss ≥ 5% from baseline to week 36 | 36 weeks
  To determine whether AZD6234 is superior to placebo in participants with weight loss ≥ 5% from baseline
Weight loss ≥ 10% from baseline to week 36 | 36 weeks
  To determine whether AZD6234 is superior to placebo in participants with weight loss ≥ 10% from baseline
Percent change in body weight from baseline to week 36 | 36 weeks
  To determine whether AZD6234 is superior to placebo for weight loss
Absolute change in body weight (kg) from baseline to week 26 and week 36 | week 26 and week 36
  To determine whether AZD6234 is superior to placebo for absolute weight loss
AZD6234 plasma concentrations | Week 43
  To characterise the PK of AZD6234

CONTACTS AND LOCATIONS:
Locations (39):
- United States (22):
  - Research Site, Mobile, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Long Beach, California
  - Research Site, Hialeah, Florida
  - Research Site, Largo, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Woodstock, Georgia
  - Research Site, Indianapolis, Indiana
  - Research Site, Lutherville-Timonium, Maryland
  - Research Site, Gulfport, Mississippi
  - Research Site, Ridgeland, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Portsmouth, New Hampshire
  - Research Site, Statesville, North Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Port Arthur, Texas
  - Research Site, San Antonio, Texas
- Australia (4):
  - Research Site, Heidelberg
  - Research Site, Maroochydore
  - Research Site, Maroubra
  - Research Site, Merewether
- Canada (6):
  - Research Site, Hamilton, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Stouffville, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
- United Kingdom (4):
  - Research Site, Hull
  - Research Site, Leicester
  - Research Site, Penarth
  - Research Site, Rotherham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/